CLINICAL TRIAL: NCT05564481
Title: Optimizing Technology Uptake and Use in Hard to Reach Adolescents With Type 1 Diabetes
Brief Title: Research on Optimizing the Use of Technology With Education
Acronym: ROUTE-T1D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Randi Streisand, Chief of Psych/Behavioral Hlth, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00016314
Record Dates: First submitted 2022-08-26; First posted 2022-10-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes; Continuous Glucose Monitoring; Behavioral Intervention; Parent-Child Relations
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: wait-list control; all participants receive intervention- randomized to start immediately or 6 months after CGM start
Who Masked: Outcomes Assessor
Masking Description: a research assistant blind to condition of participant will complete outcome assessments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immediate intervention (Experimental): Participants randomized to the immediate intervention group will participate in 3 video-conferencing sessions with a Certified Diabetes Care and Education Specialist (CDCES) interventionist and connect with a peer parent consultant immediately post randomization (expected intervention duration: 3 months).
  Interventions: Behavioral: diabetes education and parent coaching support
- Wait-list/delayed intervention (Active Comparator): Participants randomized to the delayed intervention group will receive no intervention for 6 months post-randomization; after the 6-month follow-up period, the delayed intervention group also will participate in 3 video conferencing sessions with a CDCES interventionist and connect with a peer parent consultant (expected intervention duration: 3 months).
  Interventions: Behavioral: diabetes education and parent coaching support

INTERVENTIONS:
Behavioral: diabetes education and parent coaching support — Intervention sessions will include parent/child discussion about barriers to CGM use, review of CGM data, problem solving, and working as a team.

SUMMARY:
Consistent use of continuous glucose monitors (CGM) has the potential to improve glycemic control and related type 1 diabetes (T1D) health outcomes, however young adolescents with T1D are the least likely age group to begin and sustain use of CGM. The proposed study will conduct a feasibility trial of a behavioral intervention designed to optimize use of CGM in adolescents specifically targeting underrepresented populations in diabetes technology research.

DETAILED DESCRIPTION:
Young adolescents (ages 10-15) with type 1 diabetes (T1D) are at high risk for deterioration of glycemic control and relatedly poor overall T1D self-management. Continuous glucose monitors (CGM) provide real-time indicators of glucose levels and alert users to hypoglycemia and hyperglycemia. Consistent, informed use of CGM has the potential to improve glycemic control and related T1D health outcomes. However, adolescents with T1D are the least likely age group to utilize CGM and significant health disparities exist in access to and use of CGM among youth from racial and ethnic minority backgrounds and youth with public insurance. Adolescent CGM users also continue to evidence A1c levels above recommended targets, potentially due challenges related to perceived CGM burden and related family functioning. Novel, developmentally targeted interventions delivered early in adolescence could promote optimal uptake and use of CGM and reduce psychosocial barriers to sustained use but must be evaluated in rigorous pilot trials that attend to health disparities. The current study proposes to evaluate an innovative behavioral intervention that utilizes certified diabetes care and education specialists (CDCES) to teach problem-solving and communication skills around CGM data and use, targeting adolescent-parent T1D interactions related to glucose data, individualized CGM challenges, and weekly adolescent-parent joint review of CGM reports. The intervention also addresses HCP knowledge of health disparities in diabetes technology through interactive education, and boosts family support through connection with peer parent consultants. This study aims to evaluate the preliminary efficacy of the behavioral intervention to enhance CGM use and resulting T1D health outcomes. Sixty adolescents and their parents will be recruited for this pilot randomized trial, randomly assigned to either an immediate intervention group or a delayed intervention group serving as a standard care comparison. Intervention content will be delivered via 3 telemedicine sessions with adolescents and a parent and supported by connection with a peer parent consultant. Medical and psychosocial data (including A1c, CGM indicators, CGM burdens and benefits, diabetes distress, and diabetes-related family conflict) will be collected from adolescents and a parent at baseline and three follow-up time points across the first year after CGM initiation. The investigators will employ quantitative and qualitative analyses to evaluate intervention feasibility, acceptability, and impact. Enhancing CGM access and use at this key developmental juncture provides an excellent opportunity for tailored support and problem-solving, resulting in potentially lasting improvement in diabetes self-management. Results of this pilot trial will directly inform a multi-site randomized clinical trial to evaluate efficacy, with the long term goal of identifying effective behavioral strategies that can be integrated into routine diabetes education and care.

ELIGIBILITY:
Inclusion Criteria:

* 10-15 years old
* Type 1 diabetes
* Type 1 diabetes diagnosis ≥ 6 months \
* Starting a continuous glucose monitor for the first time or restarting after ≥ 1 year

Exclusion Criteria:

* Younger than 10, older than 15
* Diagnosed less than 6 months
* Already using CGM or has used within last year
* Other major medical condition such as cancer, cystic fibrosis

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | Baseline
  hemoglobin A1c (HbA1c)
Glycemic control | 3 months post randomization
  hemoglobin A1c (HbA1c)
Glycemic control | 6 months post randomization
  hemoglobin A1c (HbA1c)
Glycemic control | 12 months post randomization
  hemoglobin A1c (HbA1c)
glycemic variability | Baseline
  Using 14-30 days of CGM data
glycemic variability | 3 months post randomization
  Using 14-30 days of CGM data
glycemic variability | 6 months post randomization
  Using 14-30 days of CGM data
glycemic variability | 12 months post randomization
  Using 14-30 days of CGM data

SECONDARY OUTCOMES:
Family Conflict | Baseline
  The Diabetes Family Conflict Scale-Revised Scored 19-57 where a higher score indicates higher family conflict
Family Conflict | 3 months post randomization
  The Diabetes Family Conflict Scale-Revised Scored 19-57 where a higher score indicates higher family conflict
Family Conflict | 6 months post randomization
  The Diabetes Family Conflict Scale-Revised Scored 19-57 where a higher score indicates higher family conflict
Family Conflict | 12 months post randomization
  The Diabetes Family Conflict Scale-Revised Scored 19-57 where a higher score indicates higher family conflict
Diabetes Distress | Baseline
  Problem Areas in Diabetes scales (PAID) Scored 14-84 where higher scores indicate higher distress
Diabetes Distress | 3 months post randomization
  Problem Areas in Diabetes scales (PAID) Scored 14-84 where higher scores indicate higher distress
Diabetes Distress | 6 months post randomization
  Problem Areas in Diabetes scales (PAID) Scored 14-84 where higher scores indicate higher distress
Diabetes Distress | 12 months post randomization
  Problem Areas in Diabetes scales (PAID) Scored 14-84 where higher scores indicate higher distress
CGM benefits and burdens | Baseline
  Continuous glucose monitoring (CGM) Burdens and Benefits as assessed by The BenCGM and BurCGM
CGM benefits and burdens | 3 months post randomization
  Continuous glucose monitoring (CGM) Burdens and Benefits as assessed by The BenCGM and BurCGM
CGM benefits and burdens | 6 months post randomization
  Continuous glucose monitoring (CGM) Burdens and Benefits as assessed by The BenCGM and BurCGM
CGM benefits and burdens | 12 month post randomization
  Continuous glucose monitoring (CGM) Burdens and Benefits as assessed by The BenCGM and BurCGM
CGM use | Baseline
  Indicators of CGM use, including mean days work per week, will be evaluated to measure sustained use of CGM.
CGM use | 3 months post randomization
  Indicators of CGM use, including mean days work per week, will be evaluated to measure sustained use of CGM.
CGM use | 6 months post randomization
  Indicators of CGM use, including mean days work per week, will be evaluated to measure sustained use of CGM.
CGM use | 12 months post randomization
  Indicators of CGM use, including mean days work per week, will be evaluated to measure sustained use of CGM.
Diabetes self-management | Baseline
  The Diabetes Management Questionnaire (DMQ)-a self- and parent-report measure assessing the frequency of engagement in diabetes care behaviors (e.g. BG monitoring, adjusting behavior to specific situations) over the past month.
  Scored 0-100 with higher scores indicating higher adherence to diabetes management
Diabetes self-management | 3 months post randomization
  The Diabetes Management Questionnaire (DMQ)-a self- and parent-report measure assessing the frequency of engagement in diabetes care behaviors (e.g. BG monitoring, adjusting behavior to specific situations) over the past month.
  Scored 0-100 with higher scores indicating higher adherence to diabetes management
Diabetes self-management | 6 months post randomization
  The Diabetes Management Questionnaire (DMQ)-a self- and parent-report measure assessing the frequency of engagement in diabetes care behaviors (e.g. BG monitoring, adjusting behavior to specific situations) over the past month.
  Scored 0-100 with higher scores indicating higher adherence to diabetes management
Diabetes self-management | 12 months post randomization
  The Diabetes Management Questionnaire (DMQ)-a self- and parent-report measure assessing the frequency of engagement in diabetes care behaviors (e.g. BG monitoring, adjusting behavior to specific situations) over the past month.
  Scored 0-100 with higher scores indicating higher adherence to diabetes management

CONTACTS AND LOCATIONS:
Overall Officials: Randi Streisand, PhD, Principal Investigator — Children's National Hosptial
Locations (1):
- Children's National Research Institute, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No